CLINICAL TRIAL: NCT04709783
Title: Implementing 3-Step Workout for Life to Improve ADL Outcome in Home Health
Brief Title: Implementing 3-Step Workout for Life in Home Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to recruit sufficient participants during the funding period.
Sponsor: University of Florida (Other)
Collaborators: American Occupational Therapy Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB202001011
Record Dates: First submitted 2021-01-07; First posted 2021-01-14 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Frailty; Disability or Chronic Disease Leading to Disablement
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation Arm (Experimental): Participants will receive the 3-Step Workout for Life program and other rehabilitation services based on the plan of care.
  Interventions: Other: 3-Step Workout for Life

INTERVENTIONS:
Other: 3-Step Workout for Life — Participants will receive the modified 3-step Workout for Life program given by their physical therapy or occupational therapy providers. The program includes single-joint and multiple joint progressive resistance exercise and activities of daily living exercise. During the resistance exercise sessions, participants will use resistance tubing to strengthen major muscle groups of the upper extremity and/or lower extremity. During the activities of daily living exercise, participants will practice activities of daily living that they experience difficulty. The intervention volume, duration, and frequency will be modified to enhance practicality in a home health care setting over the implementation phase. In addition to the 3-Step Workout for Life exercise, participants may also receive other routine rehabilitation treatment determined and provided by their therapists to facilitate their functional recovery.

SUMMARY:
The purpose of this project is to study how to adapt and implement the 3-Step Workout for Life program in a local home health agency. A series of learning cycles will be conducted to adjust the treatment dose and delivery mode. The specific aim is to evaluate the implementation-related clinical and patient outcomes.

DETAILED DESCRIPTION:
Medicare beneficiaries admitted to home health agencies are often in frail status with decreased muscle strength and difficulty in performing activities of daily living. The purpose of the proposed research is to study how to adapt and implement the 3-Step Workout for Life program by the physical therapy and occupational therapy practitioners in a local home health agency. A series of learning cycles will be conducted to adjust the treatment dose and delivery mode, so that the program can be implemented at low cost but remains effective in improving self-care ability for Medicare beneficiaries. The specific aim is to evaluate the implementation-related clinical and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* is a Medicare beneficiary
* admitted to the partnered home health agency
* show or experience muscle weakness
* demonstrate functional limitation on at least one of the OASIS self-care items

Exclusion Criteria:

* has an acute fracture with surgical or weight-bearing restrictions
* has elective joint replacement surgery
* has a lower extremity amputation
* is receiving active treatment for cancer diagnosis
* has on-going dialysis treatment
* had acute cardiac surgery
* with acute stroke or neurologic disorder that limits motor movements
* in terminal stages of congestive heart failure
* has been referred to hospice care
* has severe cognitive deficits limiting verbal communication
* has significant medical complications that preclude safe participation in resistance exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiung-ju Liu, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu CJ, Jones LY, Formyduval A RM, Clark DO. Task-Oriented Exercise to Reduce Activities of Daily Living Disability in Vulnerable Older Adults: A Feasibility Study of the 3-Step Workout for Life. J Aging Phys Act. 2016 Jul;24(3):384-92. doi: 10.1123/japa.2015-0070. Epub 2015 Nov 19. PMID 26583695
- [Background] Liu CJ, Xu H, Keith NR, Clark DO. Promoting ADL independence in vulnerable, community-dwelling older adults: a pilot RCT comparing 3-Step Workout for Life versus resistance exercise. Clin Interv Aging. 2017 Jul 19;12:1141-1149. doi: 10.2147/CIA.S136678. eCollection 2017. PMID 28769559
- [Background] Liu CJ, Donovan J, Wolford CL. Feasibility of staff-led 3-Step Workout for Life to reduce late-life activities of daily living disability: a community-based translational study. Int J Rehabil Res. 2020 Jun;43(2):141-147. doi: 10.1097/MRR.0000000000000396. PMID 32073464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two offices of a local home health agency. The home health therapy staff screened and referred eligible home health patients between April 2022 and March 2023. The first eligible participant was enrolled on May 26, 2022, and the last was enrolled in February 2023.
Pre-assignment Details: Of 10 enrolled patients, all received the modified 3-Step Workout for Life program.
Groups:
- Implementation Arm: Participants received the modified 3-Step Workout for Life program and other rehabilitation services based on the plan of care.
  3-Step Workout for Life: Participants received the 3-step Workout for Life program given by their physical therapy or occupational therapy providers. The program includes single-joint and multiple joint progressive resistance exercise and activities of daily living exercise training. During the resistance exercise sessions, participants will use resistance tubing to strengthen major muscle groups of the upper extremity and lower extremity. During the activities of daily living exercise, participants will practice activities of daily living that they experience difficulty. The intervention volume, duration, and frequency will be modified to enhance practicality in a home health care setting over the implementation phase. In addition to the 3-Step Workout for Life, participants may also receive other routine rehabilitation treatment determined and provided by their therapists to facilitate their functional recovery.
Period: Overall Study
Arm/Group | Implementation Arm
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Implementation Arm: Participants will receive the modified 3-Step Workout for Life program and other rehabilitation services based on the plan of care.
  3-Step Workout for Life: Participants will receive the modified 3-step Workout for Life program given by their physical therapy or occupational therapy providers. The program includes single-joint and multiple joint progressive resistance exercise and activities of daily living exercise. During the resistance exercise sessions, participants will use resistance tubing to strengthen major muscle groups of the upper extremity and/or lower extremity. During the activities of daily living exercise, participants will practice activities of daily living that they experience difficulty. The intervention volume, duration, and frequency will be modified to enhance practicality in a home health care setting over the implementation phase. In addition to the 3-Step Workout for Life exercise, participants may also receive other routine rehabilitation treatment determined and provided by their therapists to facilitate their functional recovery.
Arm/Group | Implementation Arm
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.8 (6.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Ratio OASIS (Outcome and Assessment Information Set): Self-care and mobility [Mean (Standard Deviation); unit: Ratio] — The self-care and mobility measures are obtained from the OASIS (Outcome and Assessment Information Set). Each measure is indicated by a ratio score. A ratio score is calculated as the sum of attempted activity scores divided by the maximal total score of attempted activities. Each ratio score ranges from 0.17 to 1. A higher ratio score means a higher ability to independently perform self-care or mobility tasks.
  Ratio
    Self-care | .65 (.08)
    Mobility | .63 (.1)
Activity Measure of Post-Acute Care-Home Health Version [Mean (Standard Deviation); unit: T-scale score] — To assess the degree of difficulty in performing tasks in three domains: basic mobility, daily activities, and cognitive tasks. The raw score under each domain is then converted to a standardized T-scale score. According to the testing manual, the T-scale score range for basic mobility is from 30.36 to 70.71, for daily activities is from 22.45 to 61.92, and for applied cognition is from 9.89 to 49.40. A higher score indicates a better mobility, self-care, or functional cognition performance. The manual does not provide information on clinically relevant thresholds or mean/SD of the T-scale.
  T-scale score
    Basic Mobility Domain | 50.15 (6.52)
    Daily Activity Domain | 49.53 (9.35)
    Applied Cognitive Domain | 44.35 (6.92)
European Quality of Life 5 Dimensions [Mean (Standard Deviation); unit: units on a scale] — European Quality of Life 5 Dimensions (EuroQol) is a self-reported quality of life measure, which includes two parts.
  The EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) evaluates health status across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. An index score ranges from -0.59 (worst health) to 1 (best health).
  The EuroQol-visual analogue scales (EQ-VA) records the patient's self-rated health on a vertical visual analog scale ranging from 0 to 100. A higher score indicates better self-perceived health status.
  units on a scale
    EQ-5D-5L | .49 (.27)
    EQ-VA | 57 (29.08)

OUTCOME MEASURES:

1. Primary Outcome: Ratio OASIS (Outcome and Assessment Information Set) Items: Self-care
Description: The self-care measure is from the OASIS. It evaluates the degree of independence in seven activities: eating, oral hygiene, toileting hygiene, upper body dressing, lower body dressing, showering/bathing, and putting on/removing footwear. Each activity is scored on a six-point Likert scale ranging from 1 (totally dependent) to 6 (totally independent). A ratio score is calculated as the sum of attempted activity scores divided by the maximal total score of attempted activities. For example, if the participant is dependent on all six self-care activities, the ratio score of this participant is 0.17 (= 7*1/7*6). The ratio score of OASIS self-care ranges from 0.17 (totally dependent on all self-care activities) to 1 (totally independent of all self-care activities). A higher ratio score means a higher ability to perform self-care.
Time Frame: Discharge, on average 2 months
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Implementation Arm
Number analyzed (Participants) | 9
Ratio | 0.93 (0.14)
Statistical Analysis 1: Comparison: Implementation Arm; Test type: Other — One group pre-post test; p = .01, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.67

2. Secondary Outcome: Ratio OASIS (Outcome and Assessment Information Set) Items: Mobility
Description: The mobility measure from OASIS evaluates the degree of independence in 17 mobility activities, such as roll left and right or sit to lying. Each activity is scored on a six-point Likert scale ranging from 1 (totally dependent) to 6 (totally independent). A ratio score is calculated as the sum of attempted activity scores divided by the maximal total score of attempted activities. For example, if the participant is dependent on all 17 mobility activities, the ratio score of this participant is 0.17= 0.06 (17*1/17*6). The ratio score of OASIS mobility ranges from 0.17 (totally dependent on all mobility activities) to 1 (totally independent of all mobility activities). A higher ratio score means a higher ability to perform mobility tasks independently.
Time Frame: Discharge, on average 2 months
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Implementation Arm
Number analyzed (Participants) | 9
Ratio | 0.89 (0.19)
Statistical Analysis 1: Comparison: Implementation Arm; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.49

3. Secondary Outcome: EuroQoL (European Quality of Life)
Description: EuroQoL is a self-reported quality of life measure. The EQ-5D-5L (EuroQol-5 Dimensions-5 Levels) evaluates health status across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. An index score ranges from -0.59 (worst health) to 1 (best health).
  The EQ VAS (EuroQol_visual analogue scale) records the patient's self-rated health on a vertical visual analog scale ranging from 0 to 100. A higher score indicates better self-perceived health status.
Time Frame: Discharge, on average 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implementation Arm
Number analyzed (Participants) | 10
score on a scale
  EQ-5D-5L | 0.68 (.22)
  EQ-VAS | 64.5 (22.29)
Statistical Analysis 1: Comparison: Implementation Arm; Test type: Other; p = 0.07, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.84

4. Secondary Outcome: Activity Measure of Post-Acute Care-Home Health Version
Description: The measure evaluates the degree of difficulty in performing tasks in three domains: basic mobility, daily activities, and cognitive tasks. The raw score under each domain is then converted to a standardized T-scale score. According to the testing manual, the T-scale score range for basic mobility is from 30.36 to 70.71, for daily activities is from 22.45 to 61.92, and for applied cognition is from 9.89 to 49.40. A higher score indicates a better mobility, daily activities, or functional cognition performance. The manual does not provide information on clinically relevant thresholds or mean/SD of the T-scale.
Time Frame: Discharge, on average 2 months
Measure: Mean (Standard Deviation); unit: T-scale score
Arm/Group | Implementation Arm
Number analyzed (Participants) | 10
T-scale score
  Basic Mobility Domain | 55.77 (7.64)
  Daily Activity Domain | 54.96 (7.22)
  Applied Cognitive Domain | 45.44 (5.98)
Statistical Analysis 1: Comparison: Implementation Arm; Test type: Other; p = 0.02, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -2.37

ADVERSE EVENTS:
Time Frame: Two months
Description: The study therapy staff will check and record the adverse events of each patient and document the events. An "adverse event" is any untoward medical occurrence in a patient, not necessarily have a causal relationship with the study. A "serious adverse event" is any untoward medical occurrence that: a) results in death, b) is life-threatening, c) requires hospitalization or prolongation of existing hospitalization, or d) results in persistent or significant disability or incapacity.
Arm/Group | Implementation Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implementation Arm (N=10)
Anticipated adverse event (Musculoskeletal and connective tissue disorders) | 6 (6) — Muscle soreness and/or joint pain
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Fall

LIMITATIONS AND CAVEATS:
Not able to meet the recruitment goal within the funding period, leading to small number of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT04709783/Prot_SAP_000.pdf